CLINICAL TRIAL: NCT03720275
Title: Evaluation of a New Diagnostic Approach to Familial Amyloid Neuropathy by Mutation of the TTR Gene in a Population of Idiopathic Chronic Neuropathies
Brief Title: Early and Systematic Screening in Chronic Neuropathy
Acronym: TTR-FAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: University of Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2016/35
Record Dates: First submitted 2018-10-12; First posted 2018-10-25 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Amyloid Neuropathies, Familial
Keywords: proportion, TTR-FAP, study, neuropathy
MeSH Terms: conditions — Amyloid Neuropathies, Familial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with chronic neuropathy of unknown aetiology (Experimental): For the 130 patients with chronic neuropathy of unknown aetiology, the diagnosis of TTR-FAP will be performed using standard procedures following international recommendations, requiring genetic analysis of the TTR gene.
  Interventions: Genetic: Systematic screening of TTR mutations

INTERVENTIONS:
Genetic: Systematic screening of TTR mutations — The diagnosis of TTR-FAP requires genetic analysis using direct sequencing of TTR gene.The diagnosis of TTR-FAP will be performed using standard procedures following international recommendations, requiring genetic analysis of the TTR gene.

SUMMARY:
TTR-FAP is a rare disabling inherited disorder that predominantly affects the peripheral nervous system and the heart. Due to an important phenotypic and genetic heterogeneity, the diagnosis is often delayed, preventing therefore early onset treatment. Our project is to evaluate the prevalence of TTR-FAP in a series of 130 patients with from chronic neuropathy of undetermined aetiology through a systematic screening of TTR mutations.

DETAILED DESCRIPTION:
Transthyretin familial amyloid polyneuropathy (TTR-FAP) is an autosomal dominant disorder, highly disabling and life-threatening, resulting of transthyretin (TTR) gene mutation. Clinically, TTR FAP is characterized by progressive sensorimotor and dysautonomic neuropathy, usually fatal within a few years. The disease prevalence is highly variable, with a large genotypic and phenotypic heterogeneity. Early and accurate diagnosis remains essential to propose early treatment. New pharmacotherapies have been developed, such as Tafamidis®, and many patients can avoid liver transplant formerly considered as the only therapeutic option. The prevalence of TTR-FAP disease has been previously estimated in series of patients with severe and progressive neuropathy, frequently leading to a delayed diagnosis. TTR-FAP is also easily suspected when neuropathy is associated with cardiac symptoms or dysautonomia.

Currently, genetic testing of TTR-FAP is targeted and is only prescribed to patients in whom the first-line assessment recommended by the High Authority for Health (HAS) did not identify a cause, and on the basis of a worsening of symptoms. An early diagnosis in those cases would allow earlier treatment and monitoring. No data are available about the prevalence of TTR-FAP in populations of patients with from chronic neuropathy of unknown aetiology, through a systematic screening of TTR mutations.

The diagnosis of TTR-FAP will be performed using standard procedures following international recommendations, requiring genetic analysis of the TTR gene.

The patients with a diagnosis of TTR-FAP confirmed during this study will be seen for an additional visit in the Investigating Centre and proposed suitable follow up, treatment and care.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes presenting chronically (> 3 months):

  * neuropathy confirmed by an electroneuromyography
  * without obvious etiology (diabetes, alcohol consumption, renal insufficiency, neurotoxic substances intake, family history of diagnosed hereditary neuropathy)
  * without anomaly of the following biological examinations: fasting blood glucose, blood count, gamma-glutamyl transferases, average cell volume, transaminases, serum creatinine clearance, C-reactive protein, TSH
* Aged 18 to 90 years Patients giving their free and informed consent to participate, after research information

Exclusion Criteria:

* People placed under the protection of justice.
* Patients who are not affiliated or who are not beneficiaries of a social security scheme
* Patients with chronic neuropathy related to a known etiology

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2020-05-27 (Actual); Study Completion 2021-12-23 (Actual)

PRIMARY OUTCOMES:
Diagnosis of TTR-FAP | Genetic analyzes will be performed every three months from the first inclusion
  Proportion of TTR-FAP in the 130 patients with chronic neuropathy of unknown aetiology

SECONDARY OUTCOMES:
Age of patient at diagnosis | at the inclusion visit
History of dysautonomias | at the inclusion visit
  History of dysautonomias at the interview
Signs of dysautonomias | at the inclusion visit
  signs of dysautonomias at the interview
Weight of patient | at the inclusion visit
  weight
Height of patient | at the inclusion visit
  height
Motor deficit of the lower limbs evaluated by a subscore of the Neuropathy Impairment Scale (NIS) | at the inclusion visit
  The Motor deficit of the lower limbs will be assessed through a sub score of the Neuropathy Impairment Scale (NIS). The maximum score on the NIS scale is 244 points. The motor sub score, including the evaluation of the upper and lower limbs, is scored on 192 points. This scale allows to obtain a quantification of the clinical examination. Each item is evaluated between 0 and 4 points.
Motor deficit of the upper limbs evaluated by a subscore of the Neuropathy Impairment Scale (NIS) | at the inclusion visit
  The Motor deficit of the upper limbs will be assessed through a sub score of the Neuropathy Impairment Scale (NIS). The maximum score on the scale is 244 points. The motor sub score, including the evaluation of the upper and lower limbs, is scored on 192 points. This scale allows to obtain a quantification of the clinical examination. Each item is evaluated between 0 and 4 points.
Sensory deficit evaluated by a subscore of the Neuropathy Impairment Scale (NIS) | at the inclusion visit
  The Sensory deficit will be assessed through a sub score of the Neuropathy Impairment Scale (NIS). The maximum score on the scale is 244 points. The sensory sub score is scored on 20 points. This scale allows to obtain a quantification of the clinical examination. Each item is evaluated between 0 and 2 points.
Presence / Absence of reflexes osteo-tendinous evaluated by a subscore of the Neuropathy Impairment Scale (NIS) | at the inclusion visit
  The Presence/Absence of reflexes osteo-tendinous will be assessed through a sub score of the Neuropathy Impairment Scale (NIS). The maximum score on the scale is 88 points. The reflexes sub score is scored on 8 points. This scale allows to obtain a quantification of the clinical examination. Each item is evaluated between 0 and 2 points.
Presence of orthostatic hypotension | at the inclusion visit
  Blood pressure measurement by the nurse
Dysautonomia score | at the inclusion visit
  Score at the clinical scale assessing autonomic dysfunction according to 5 modalities: orthostatic hypotension, high digestive motor disorders, low digestive motor disorders, vesicosphincteric disorders, erectile dysfunction
Rasch-built Overall Disability Scale (RODS) score | at the inclusion visit
  Score at the RODS, a functional scale that captures daily activity and social participation limitations in patients affected by polyneuropathy (self-questionnaire)
Overall Neuropathy Limitations Scale (ONLS) score | at the inclusion visit
  The ONLS is a validated neuropathy functional scale evaluating the performance of upper and lower cells. The upper limbs sub score is scored on 5 points and the lower limbs sub score is scored on 7 points. The scale thus ranges from 0 (no disability) to 12 points (disability maximum)
Electroneuromyography findings (ENMG): axonal, demyelinating or mixed neuropathy). | at the inclusion visit

CONTACTS AND LOCATIONS:
Overall Officials: Guilhem Solé, MD, Principal Investigator — University Hospital Bordeaux, France
Locations (1):
- Reference center for neuromuscular diseases, Bordeaux, France